CLINICAL TRIAL: NCT03722030
Title: Feasibility and Acceptability of a Telehealth-Based Resistance Training Intervention for Endometrial Cancer Survivors
Brief Title: Telehealth-Based Resistance Training Intervention for Endometrial Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH); American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UW18013; P30CA014520 (NIH); NCI-2018-02257 (Registry Identifier: NCI CTRP); 2018-0953 (Other: IRB); 1R03CA230965-01A1 (NIH); A176000 (Other: UW Madison); EDUC/KINESIOLOGY (Other: UW Madison)
Record Dates: First submitted 2018-10-16; First posted 2018-10-26 (Actual); Results first posted 2020-08-11 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-06

CONDITIONS: Endometrial Cancer
Keywords: Strength Training; Resistance Training; Obesity; Sedentary
MeSH Terms: conditions — Endometrial Neoplasms; Obesity; Sedentary Behavior | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Pilot/Feasibility trial - 2 arms, one strength-training intervention vs. waitlist control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strength-Training Intervention (Experimental): Following baseline measures, participants will receive an initial in-person instructional session, instructional material and resistance training equipment, support and feedback via video coaching, mid-point assessment, and an in-person study visit to collect post study measures. Intervention will be 10 weeks, with a 5 week follow up period.
  Interventions: Other: Baseline Measures; Behavioral: Strength-Training; Other: Mid-point Measures; Other: Post-Study Measures
- Waitlist Control (Placebo Comparator): Following baseline measures, participants will provide mid-point measures, and in-person post-study measures with no 10-week strength training intervention.
  Interventions: Other: Baseline Measures; Other: Mid-point Measures; Other: Post-Study Measures

INTERVENTIONS:
Other: Baseline Measures — Accelerometer (steps), Biomarkers (finger prick for hemoglobin A1c and c-reactive protein), Anthropometrics (height, weight, waist and hip circumference), Body composition (dual-energy absorptiometry for measuring fat mass, lean mass, % body fat, visceral fat), Functional fitness test.
Behavioral: Strength-Training — 2 sessions per week (20-40 min), home-based resistance training
  Arms: Strength-Training Intervention
Other: Mid-point Measures — Accelerometer (steps)
Other: Post-Study Measures — Accelerometer (steps), Biomarkers (finger prick for hemoglobin A1c and c-reactive protein), Anthropometrics (height, weight, waist and hip circumference), Body composition (dual-energy absorptiometry for measuring fat mass, lean mass, % body fat, visceral fat), Functional fitness test.

SUMMARY:
This 2-arm pilot trial will enroll 40 participants to test the feasibility, adherence, and benefits of a home-based strength training intervention for endometrial cancer survivors relative to a wait-listed control group.

DETAILED DESCRIPTION:
Endometrial cancer survivors have an extremely high prevalence of inactivity and obesity. Inactivity and obesity are associated with poorer outcomes among survivors. Other interventions have demonstrated that walking and aerobic exercise are safe and feasible in endometrial cancer patients. However few published studies have examined strength training in endometrial cancer survivors, and these have done so only in combination with aerobic intervention (and often also dietary change) in the context of a larger multi-component intervention.

There is a critical need for data about the feasibility and benefits of strength training in this population. The investigators propose a 2-arm pilot trial of a home-based strength training intervention (vs. waitlist control) among 40 endometrial cancer survivors. The intervention will consist of (a) an initial in-person instructional session; (b) instructional materials and resistance training equipment (e.g., resistance bands) and (c) support and feedback provided via video coaching sessions. The purpose of a pilot trial is not to conduct hypothesis testing, but rather to field-test the logistical components of the study to incorporate into a larger, future study design.

The proposed trial will determine the feasibility of an at-home resistance training protocol and measurements of exercise logging, functional fitness testing, DXA, dried blood spots and questionnaire measures. Participants will be assigned either to the resistance training program (i.e., initial in-person instructional session, telephone coaching, and self-monitoring) or to a comparison arm (wait-list control).

* Aim 1: To determine the feasibility of recruiting and retaining endometrial cancer survivors to a home- based resistance training 2 sessions per week of 20-40 minutes of exercise.
* Aim 2: To determine participant satisfaction with each component of the intervention and identify opportunities for refinement of the intervention prior to testing in a larger study.
* Aim 3: To establish that functional and objective assessments are feasible and well-tolerated in enrolled participants, as assessed using the functional fitness test (FFT) battery, dual-energy x-ray absorptiometry (DXA), finger-pricks for dried blood spots and patient-reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Willing to provide written informed consent
* Willing to comply with all study procedures and be available for the duration of the study
* Fluent in spoken and written English
* Documented diagnosis of Type I, stage I-IIIc endometrial cancer within the past 5 years
* Completion of current treatment for endometrial cancer, period of time of ≥10 weeks from treatment completion to study enrollment is required

Exclusion Criteria:

* Absolute contraindications to exercise (i.e., acute myocardial infarction, severe orthopedic or musculoskeletal limitations
* Have evidence of recurrent or metastatic disease
* Are currently performing resistance training ≥2 days per week
* Report of chest pain, shortness of breath, fainting, or angina pectoris
* Have physical disability that would limit range of motion through exercises such as sitting, standing and inability to walk one block
* Plans to move from the area
* Enrolled in another clinical trial or has used of any investigational drugs, biologics, or devices within 30 days prior to randomization
* Women who are pregnant or breast-feeding
* Not suitable for study participation due to other reasons at the discretion of the investigator

Ages: 18 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2020-03-14 (Actual); Study Completion 2020-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Cadmus-Bertram, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Carbone Cancer Center, Madison, Wisconsin, United States

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/

RESULTS

PARTICIPANT FLOW:
Groups:
- Strength-Training Intervention: Following baseline measures, participants will receive an initial in-person instructional session, instructional material and resistance training equipment, support and feedback via video coaching, mid-point assessment, and an in-person study visit to collect post study measures. Intervention will be 10 weeks, with 5 week follow up period.
  Baseline Measures: Accelerometer (steps), Biomarkers (finger prick for hemoglobin A1c and c-reactive protein), Anthropometrics (height, weight, waist and hip circumference), Body composition (dual-energy absorptiometry for measuring fat mass, lean mass, % body fat, visceral fat), Functional fitness test.
  Strength-Training: 2 sessions per week (20-40 min), home-based resistance training
  Mid-point Measures: Accelerometer (steps)
  Post-Study Measures: Accelerometer (steps), Biomarkers (finger prick for hemoglobin A1c and c-reactive protein), Anthropometrics (height, weight, waist and hip circumference), Body composition (dual-energy x-ray absorptiometry)
Period: Overall Study
Arm/Group | Strength-Training Intervention | Waitlist Control
Started | 20 | 20
Completed | 19 | 20
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Strength-Training Intervention: Following baseline measures, participants will receive an initial in-person instructional session, instructional material and resistance training equipment, support and feedback via video coaching, mid-point assessment, and an in-person study visit to collect post study measures. Intervention will be 10 weeks, with 5 week follow up period.
- Total: Total of all reporting groups
Arm/Group | Strength-Training Intervention | Waitlist Control | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.9 (9.6) | 60.9 (8.0) | 60.9 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 20 | 20 | 40
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 20 | 19 | 39
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 42.2 (19.5) | 37.9 (8.6) | 39.9 (15.2)
Married or Partnered [Count of Participants; unit: Participants] | 15 | 13 | 28
Education [Count of Participants; unit: Participants]
  High school graduate or less | 1 | 2 | 3
  Trade school / some college | 7 | 6 | 13
  College graduate | 6 | 8 | 14
  Post-graduate degree | 6 | 4 | 10
Percentage Total Body Fat [Mean (Standard Deviation); unit: percent body fat] — Measured by Dual-energy X-ray absorptiometry (DXA)
  percent body fat | 51.6 (5.0) | 50.4 (6.8) | 51.2 (6.0)
Waist Circumference [Mean (Standard Deviation); unit: centimeters] | 107.9 (16.9) | 105.5 (15.2) | 106.8 (16.0)
Hip Circumference [Mean (Standard Deviation); unit: centimeters] | 130.2 (18.4) | 129.2 (19.4) | 129.7 (18.7)
Waist-to-Hip Ratio [Mean (Standard Deviation); unit: waist-to-hip circumference ratio] | 0.82 (0.04) | 0.83 (0.07) | 0.83 (0.06)
Tumor Stage At Diagnosis [Count of Participants; unit: Participants] — Staging by pathologist per the World Health Organization Classification of Tumours of the Female Genital Tract, published in 2020
  Participants
    Stage 1 | 15 | 18 | 33
    Stage 2 | 2 | 0 | 2
    Stage 3 | 3 | 2 | 5
Treatment [Count of Participants; unit: Participants]
  No treatment beyond surgery | 14 | 16 | 30
  Radiation alone | 2 | 1 | 3
  Chemotherapy alone | 0 | 3 | 3
  Chemotherapy and Radiation | 4 | 0 | 4
Time since diagnosis [Mean (Standard Deviation); unit: years] | 2.8 (1.2) | 3.0 (1.3) | 2.9 (1.2)
Time since surgery [Mean (Standard Deviation); unit: years] | 2.7 (1.4) | 3.0 (1.3) | 2.8 (1.3)

OUTCOME MEASURES:

1. Primary Outcome: Feasibility - Number of Participants Recruited
Description: The feasibility of recruiting endometrial cancer survivors to a home-based resistance training; 2 sessions per week of 20-40 minutes of exercise. This will be measured by the number of participants recruited. The goal is 40 participants.
Time Frame: up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Strength-Training Intervention | Waitlist Control
Number analyzed (Participants) | 20 | 20
Participants | 20 | 20

2. Primary Outcome: Number of Participants Who Completed 100% of the Prescribed Exercises
Description: Compliance/adherence will be measured via detailed exercise logs. A participant needs to complete at least 50% of the prescribed exercises in a session to be considered adherent to the session.
Time Frame: up to 20 weeks from beginning of intervention
Population: Waitlist control group was not included in adherence measures as they did not receive exercises until final measures were completed.
Measure: Count of Participants; unit: Participants
Arm/Group | Strength-Training Intervention | Waitlist Control
Number analyzed (Participants) | 19 | 0
Participants | 17 | 0

3. Primary Outcome: Number of Participants With Adverse Events
Description: The primary safety endpoint will be total number of adverse events over the duration of the intervention.
Time Frame: up to 20 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Strength-Training Intervention | Waitlist Control
Number analyzed (Participants) | 19 | 20
Participants | 0 | 0

4. Secondary Outcome: Number of Participants Reporting "Very" or "Extremely" Satisfied With Intervention
Description: Participants will complete semi-structured qualitative interviews with the study coordinator. Interviews will be recorded, transcribed and coded to identify content themes. These interviews will be used to collect qualitative information and overall satisfaction with the intervention, as well as areas to improve with future interventions and barriers to participation.
Time Frame: At final visit - up to 20 weeks
Population: Satisfaction was only collected for the strength training intervention. Sixteen participants completed the end of study satisfaction survey upon which this metric was based.
Measure: Count of Participants; unit: Participants
Arm/Group | Strength-Training Intervention | Waitlist Control
Number analyzed (Participants) | 16 | 0
Participants | 16 |

5. Secondary Outcome: Change in Hemoglobin A1c From Baseline
Description: Baseline and post-study blood biomarkers to assess Hemoglobin A1c will be collected and reported in a table as a change from baseline.
Time Frame: baseline and 10 weeks
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Strength-Training Intervention | Waitlist Control
Number analyzed (Participants) | 20 | 20
ng/mL | 4.7 (8.4) | 3.2 (5.9)

6. Secondary Outcome: Change in C-Reactive Protein From Baseline
Description: Baseline and post-study blood biomarkers to assess c-reactive protein will be collected and reported in a table as a change from baseline.
Time Frame: baseline and 10 weeks
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Strength-Training Intervention | Waitlist Control
Number analyzed (Participants) | 20 | 20
ng/mL | 222.1 (538.3) | 108.6 (400.9)

7. Secondary Outcome: Change in Lean Muscle Mass From Baseline
Description: Baseline and post-study lean muscle mass will be assessed using dual-energy absorptiometry (DXA) using the enCORE Lunar iDXA software suite (GE Healthcare, Little Chalfont, UK). Data will be reported in a table as change from baseline.
Time Frame: baseline and 10 weeks
Measure: Mean (Standard Deviation); unit: pounds muscle
Arm/Group | Strength-Training Intervention | Waitlist Control
Number analyzed (Participants) | 20 | 20
pounds muscle | 1.0 (2.6) | -0.7 (3.3)

8. Secondary Outcome: Change in Fat Mass From Baseline
Description: Baseline and post-study fat mass will be assessed using dual-energy absorptiometry (DXA) utilizing the enCORE Lunar iDXA software suite (GE Healthcare, Little Chalfont, UK). Data will be reported in a table as change from baseline.
Time Frame: baseline and 10 weeks
Population: Absolution change in fat mass was not reported, instead percent fat change was reported to standardize for total body mass allowing for easier interpretation across individuals.
Arm/Group | Strength-Training Intervention | Waitlist Control
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Change in Visceral Fat Mass From Baseline
Description: Baseline and post-study visceral fat mass will be assessed using dual-energy absorptiometry (DXA) utilizing the enCORE Lunar iDXA software suite (GE Healthcare, Little Chalfont, UK). Data will be reported in a table as change from baseline.
Time Frame: up to 20 weeks
Population: Visceral fat mass was not measured for all scans on each participant, therefore due to the amount of missing data, the change in visceral fat mass could not be measured.
Arm/Group | Strength-Training Intervention | Waitlist Control
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Change in Total Percent Body Fat From Baseline
Description: Baseline and post-study % body fat will be assessed using dual-energy absorptiometry (DXA) utilizing the enCORE Lunar iDXA software suite (GE Healthcare, Little Chalfont, UK). Data will be reported in a table as change from baseline.
Time Frame: baseline and 10 weeks
Measure: Mean (Standard Deviation); unit: body fat percent
Arm/Group | Strength-Training Intervention | Waitlist Control
Number analyzed (Participants) | 20 | 20
body fat percent | -0.6 (0.9) | -0.3 (1.5)

11. Secondary Outcome: Change in Number of Arm Curls Performed From Baseline
Description: Arm curls are part of the functional fitness test (FFT); a battery of tests measuring strength, flexibility, fitness, body composition, and agility. These tests will be performed at baseline and post-study time points. Data will be reported in a table as change from baseline.
  The 30 second arm curl assesses the strength of the upper body, where participants hold a 5 pound dumbbell in a seated position, and they will have 30 seconds to curl their arm and extend it as many times as possible within the time frame.
Time Frame: baseline and 10 weeks
Measure: Mean (Standard Deviation); unit: repetitions
Arm/Group | Strength-Training Intervention | Waitlist Control
Number analyzed (Participants) | 20 | 20
repetitions | 4.9 (3.7) | 2.2 (2.0)

12. Secondary Outcome: Change in Number of Sit to Stand Repetitions Performed From Baseline
Description: The 30 second chair stand is part of the functional fitness test (FFT); a battery of tests measuring strength, flexibility, fitness, body composition, and agility. This test will be performed at baseline and post-study time points. Data will be reported in a table as change from baseline.
  The 30 second chair stand assesses the strength of the lower body. Each person will have 30 seconds to stand up and sit down from a chair as many times as possible within the time frame.
Time Frame: baseline and 10 weeks
Measure: Mean (Standard Deviation); unit: repetitions
Arm/Group | Strength-Training Intervention | Waitlist Control
Number analyzed (Participants) | 20 | 20
repetitions | 3.3 (3.5) | 0.3 (2.4)

13. Secondary Outcome: Change in Handgrip Weight From Baseline
Description: Handgrip is part of the functional fitness test (FFT); a battery of tests measuring strength, flexibility, fitness, body composition, and agility. This test will be performed at baseline and post-study time points. Data will be reported in a table as change from baseline.
  [can you describe this test? I do not see it in the protocol]
Time Frame: baseline and 10 weeks
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Strength-Training Intervention | Waitlist Control
Number analyzed (Participants) | 20 | 20
kilograms | 0.7 (2.2) | -0.4 (2.1)

14. Secondary Outcome: Change in Sit and Reach Distance From Baseline
Description: The chair sit and reach test is part of the functional fitness test (FFT); a battery of tests measuring strength, flexibility, fitness, body composition, and agility. This test will be performed at baseline and post-study time points. Data will be reported in a table as change from baseline.
  The chair sit and reach assesses lower body flexibility where the participant will sit in a chair, extend one leg in front of them and flex at the waist, reaching toward their toes, the measure is the distance between their toes and fingers.
Time Frame: baseline and 10 weeks
Measure: Mean (Standard Deviation); unit: inches
Arm/Group | Strength-Training Intervention | Waitlist Control
Number analyzed (Participants) | 20 | 20
inches | 0.9 (2.3) | -0.5 (3.7)

15. Secondary Outcome: Change in Back Scratch Distance From Baseline
Description: The back scratch test is part of the functional fitness test (FFT); a battery of tests measuring strength, flexibility, fitness, body composition, and agility. This test will be performed at baseline and post-study time points. Data will be reported in a table as change from baseline.
  The back scratch test assesses the upper body flexibility, where the person is seated and one arm will be flexed behind the head, and the other arm will be extended behind the shoulder. The assessment measures the distance between the finger tips of both hands.
Time Frame: baseline and 10 weeks
Measure: Mean (Standard Deviation); unit: inches
Arm/Group | Strength-Training Intervention | Waitlist Control
Number analyzed (Participants) | 20 | 20
inches | 1.1 (1.7) | 0.1 (4.1)

16. Secondary Outcome: Change in 6-minute Walk Distance From Baseline
Description: The 6-minute walk test is part of the functional fitness test (FFT); a battery of tests measuring strength, flexibility, fitness, body composition, and agility. This test will be performed at baseline and post-study time points. Data will be reported in a table as change from baseline.
  The 6 minute walk test measures the total distance that a person can quickly walk on a flat hard surface within a period of 6 minutes, using a 100ft length of distance.
Time Frame: baseline and 10 weeks
Measure: Mean (Standard Deviation); unit: feet
Arm/Group | Strength-Training Intervention | Waitlist Control
Number analyzed (Participants) | 20 | 20
feet | 70.0 (89.3) | 34.9 (114)

17. Secondary Outcome: Change in 8 Foot Up and Go Time From Baseline
Description: The 8-foot-up and go test is part of the functional fitness test (FFT); a battery of tests measuring strength, flexibility, fitness, body composition, and agility. This test will be performed at baseline and post-study time points. Data will be reported in a table as change from baseline.
  The 8-foot-up and go is an assessment of speed agility and balance. The participant begins in a seated position and will be timed for the duration it takes to rise from the chair, walk as quickly as possible around a cone 8 feet away from the chair, and return to a seated position.
Time Frame: baseline and 10 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Strength-Training Intervention | Waitlist Control
Number analyzed (Participants) | 20 | 20
seconds | -0.7 (0.9) | -0.1 (1.0)

18. Secondary Outcome: FACT Scores
Description: Functional Assessment of Cancer Therapies (FACT) changes from baseline, mid-point, to post-study will be captured using the Functional Assessment of Cancer Therapies (FACT) questionnaire including the Endometrial subscale (FACT-En). The FACT assessment measures physical, social/family, and functional well-being, each on a scale of 0-28, and emotional well being on a scale of 0-24. The Endometrial component contains concerns specific to endometrial cancer such as hot/flashes, cramps, and swelling; measured on a scale of 0-64. Each of these sections will be scored for sub-scale scores and then the entire instrument will have a total composite score (0-172; the higher the score, the more quality of life improvements) and will be reported as such.
Time Frame: baseline, 5 weeks, 10 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Strength-Training Intervention | Waitlist Control
Number analyzed (Participants) | 20 | 20
score on a scale
  baseline | 146 (11.9) | 141 (21.7)
  Week 5 | 146 (13.2) | 142 (21.7)
  Week 10 | 146 (15.0) | 140 (26.1)

19. Secondary Outcome: Changes in FACT From Baseline
Description: as for outcome 18
Time Frame: baseline and 10 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Strength-Training Intervention | Waitlist Control
Number analyzed (Participants) | 20 | 20
score on a scale | -0.3 (14.0) | 0.6 (13.0)

20. Secondary Outcome: FACT-En Scores
Description: Functional Assessment of Cancer Therapies (FACT) changes from baseline, mid-point, to post-study will be captured using the Functional Assessment of Cancer Therapies (FACT) questionnaire including the Endometrial subscale (FACT-En). The Endometrial component contains concerns specific to endometrial cancer such as hot/flashes, cramps, and swelling; measured on a scale of 0-64, the higher the score, the more quality of life improvements.
Time Frame: baseline, 5 Weeks,10 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Strength-Training Intervention | Waitlist Control
Number analyzed (Participants) | 20 | 20
score on a scale
  Baseline | 55.0 (7.1) | 54.5 (7.1)
  Week 5 | 54.6 (7.2) | 54.7 (5.0)
  Week 10 | 55.0 (7.5) | 55.0 (7.0)

21. Secondary Outcome: Changes in FACT-En From Baseline
Description: as for outcome 20
Time Frame: baseline and 10 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Strength-Training Intervention | Waitlist Control
Number analyzed (Participants) | 20 | 20
score on a scale | -0.0 (5.1) | 0.4 (5.8)

22. Secondary Outcome: FACT Physical Subscale Scores
Description: Functional Assessment of Cancer Therapies (FACT) changes from baseline, mid-point, to post-study will be captured using the Functional Assessment of Cancer Therapies (FACT). The FACT assessment measures physical, social/family, emotional, and functional well-being, each on a scale of 0-28. Each of these sections will be scored for sub-scale scores; the higher the score, the more quality of life improvements.
Time Frame: baseline, 5 weeks, 10 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Strength-Training Intervention | Waitlist Control
Number analyzed (Participants) | 20 | 20
score on a scale
  Baseline | 24.4 (2.3) | 24.0 (3.4)
  Week 5 | 24.5 (2.9) | 23.9 (4.3)
  Week 10 | 24.8 (2.9) | 24.5 (4.5)

23. Secondary Outcome: FACT Social Subscale Scores
Description: as for outcome 22
Time Frame: baseline, 5 weeks, 10 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Strength-Training Intervention | Waitlist Control
Number analyzed (Participants) | 20 | 20
score on a scale
  Baseline | 22.3 (3.2) | 20.6 (6.5)
  Week 5 | 22.4 (5.0) | 20.8 (6.0)
  Week 10 | 22.3 (4.8) | 19.7 (7.6)

24. Secondary Outcome: FACT Emotional Subscale Scores
Description: as for outcome 22
Time Frame: baseline, 5 weeks, 10 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Strength-Training Intervention | Waitlist Control
Number analyzed (Participants) | 20 | 20
score on a scale
  Baseline | 21.1 (2.7) | 20.4 (3.3)
  Week 5 | 21.4 (2.4) | 20.7 (3.3)
  Week 10 | 20.8 (3.8) | 20.2 (3.4)

25. Secondary Outcome: FACT Functional Subscale Scores
Description: as for outcome 22
Time Frame: baseline, 5 weeks, 10 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Strength-Training Intervention | Waitlist Control
Number analyzed (Participants) | 20 | 20
score on a scale
  Baseline | 23.0 (2.6) | 21.6 (5.0)
  Week 5 | 22.9 (3.2) | 21.7 (5.3)
  Week 10 | 23.3 (3.5) | 21.0 (6.3)

26. Secondary Outcome: Changes in FACT Subscales From Baseline
Description: as for outcome 22
Time Frame: baseline and 10 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Strength-Training Intervention | Waitlist Control
Number analyzed (Participants) | 20 | 20
score on a scale
  Physical | 0.4 (2.7) | 0.5 (2.5)
  Social | -0.0 (3.6) | -0.7 (3.8)
  Emotional | -0.4 (3.3) | -0.1 (3.0)
  Functional | 0.3 (2.8) | -0.5 (3.3)

27. Secondary Outcome: Changes in Mental Well-being From Baseline
Description: Changes in mental well-being from baseline, mid-point, and post-study (including anxiety, depression, and fatigue) will be assessed using standardized NIH-provided Patient-Reported Outcome Measurement Information System (PROMIS) measures.
  The fatigue assessment asks about self-reported systems of fatigue and tiredness, all the way up to exhaustion overall, and ask about fatigue over the past seven days. The depression assessment asks about depressive symptoms over the past seven days. The anxiety assessment asks about symptoms adjacent-to and including anxiety over the past seven days. For each of these three instruments (which comprise the mental well-being assessments) the data will be reported as change over time, specifically using the T-score (standardized mean) and the standard error.
  Each is standardized to a mean of 50 and a range of 0-100; a higher scores indicate a higher "level" of that construct, whether it's higher levels of depression, fatigue or anxiety.
Time Frame: baseline and Week 10
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Strength-Training Intervention | Waitlist Control
Number analyzed (Participants) | 20 | 20
T-score
  Anxiety | -0.3 (6.7) | 1.5 (6.6)
  Fatigue | -2.5 (7.9) | -2.0 (9.3)
  Depression | -1.8 (5.0) | -0.8 (5.4)

28. Secondary Outcome: Changes in Self-Efficacy From Baseline
Description: Self-efficacy will be assessed at baseline, mid-point, and post-study using the validated self-efficacy for exercise scale, modified for specificity to strength training.
  This instrument has 9 items, each of which is scored from 0-10, with a maximum score of 90. Higher scores indicate higher self-efficacy for exercise. These scores will be reported descriptively at each time point (baseline, mid-point, final), and will also be reported in a table as change over time.
Time Frame: Baseline and 10 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Strength-Training Intervention | Waitlist Control
Number analyzed (Participants) | 20 | 20
score on a scale | -3.4 (19.0) | -6.0 (14.7)

29. Secondary Outcome: Self-Efficacy Scores
Description: as for outcome 28
Time Frame: Baseline, 5 weeks, 10 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Strength-Training Intervention | Waitlist Control
Number analyzed (Participants) | 20 | 20
score on a scale
  baseline | 63.4 (20.4) | 63.7 (19.7)
  week 5 | 57.3 (19.0) | 58.3 (20.3)
  week 10 | 60.0 (21.3) | 57.7 (22.9)

30. Secondary Outcome: Changes in Accelerometer-Measured Physical Activity From Baseline
Description: Although aerobic and lifestyle physical activity (PA) are not a focus of the intervention, they will be assessed to determine baseline PA level and identify whether uptake of resistance training is associated with changes in other PA types. Participants will wear the ActiGraph wGT3X-BT accelerometer (ActiGraph, Pensacola, FL) for 7 days during all waking hours, at baseline, mid-point, and post-study visit. The ActiGraph is a gold standard method of objective activity assessment. Accelerometer data will be measured in total minutes of moderate to vigorous physical activity over a 7-day period.
  Light intensity is Moderate intensity is Vigorous intensity is
Time Frame: baseline and Week 10
Measure: Mean (Standard Deviation); unit: minutes per week
Arm/Group | Strength-Training Intervention | Waitlist Control
Number analyzed (Participants) | 20 | 20
minutes per week
  Light Activity | -77 (200) | 5 (306)
  Moderate Activity | -41 (72) | 5 (69)
  Vigorous Activity | 0 (3) | -2 (9)
  Moderate Vigorous Physical Activity (continuous minutes) | -41 (72) | 3 (73)
  Moderate Vigorous Physical Activity in bouts greater than 10 minutes | -30 (49) | -8 (41)

31. Secondary Outcome: Change in Steps Per Day From Baseline
Description: Although aerobic and lifestyle physical activity (PA) are not a focus of the intervention, they will be assessed to determine baseline PA level and identify whether uptake of resistance training is associated with changes in other PA types. Participants will wear the ActiGraph wGT3X-BT accelerometer (ActiGraph, Pensacola, FL) for 7 days during all waking hours, at baseline, mid-point, and post-study visit. The ActiGraph is a gold standard method of objective activity assessment. Accelerometer data will be measured in total minutes of moderate to vigorous physical activity over a 7-day period.
Time Frame: baseline and Week 10
Measure: Mean (Standard Deviation); unit: steps per day
Arm/Group | Strength-Training Intervention | Waitlist Control
Number analyzed (Participants) | 20 | 20
steps per day | -1038 (1190) | -92 (2046)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from enrollment to final data collection point, up to 15 weeks in length.
Arm/Group | Strength-Training Intervention | Waitlist Control
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-03-19): https://cdn.clinicaltrials.gov/large-docs/30/NCT03722030/Prot_SAP_000.pdf
  • Informed Consent Form (2019-05-02): https://cdn.clinicaltrials.gov/large-docs/30/NCT03722030/ICF_001.pdf